CLINICAL TRIAL: NCT03014622
Title: A Phase 3, Randomized, Double-Blind, Placebo Controlled, Multi-Center Trial to Evaluate the Efficacy and Safety of DaxibotulinumtoxinA for Injection to Treat Moderate to Severe Glabellar Lines (SAKURA-1)
Brief Title: Efficacy and Safety of DaxibotulinumtoxinA for Injection to Treat Moderate to Severe Glabellar Lines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Revance Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 1620301
Record Dates: First submitted 2016-12-22; First posted 2017-01-09 (Estimated); Results first posted 2022-07-21 (Actual); Last update posted 2022-07-21 (Actual); Status verified 2022-06

CONDITIONS: Glabellar Frown Lines
Keywords: glabellar lines, frown lines
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- DaxibotulinumtoxinA 40 units (Experimental): Biological/Vaccine: Botulinum Toxins, Type A Intramuscular injection
  Interventions: Biological: Botulinum Toxins, Type A
- Placebo (Placebo Comparator): Biological/Vaccine: Placebos Intramuscular injection
  Interventions: Biological: Placebos

INTERVENTIONS:
Biological: Botulinum Toxins, Type A — Intramuscular injection
  Other Names: DaxibotulinumtoxinA
  Arms: DaxibotulinumtoxinA 40 units
Biological: Placebos — Intramuscular injection
  Arms: Placebo

SUMMARY:
This is a safety and efficacy study of DaxibotulinumtoxinA for Injection to treat moderate to severe frown lines.

ELIGIBILITY:
Inclusion Criteria:

* Provide written informed consent including authorization to release health information
* Moderate (2) or severe (3) glabellar lines during maximum frown based on the Investigator Global Assessment Frown Wrinkle Severity (IGA-FWS) scale
* Moderate (2) or severe (3) glabellar lines during maximum frown based on the Patient Frown Wrinkle Severity (PFWS) scale
* Willing and able to follow all trial procedures, attend all scheduled visits, and successfully complete the trial

Exclusion Criteria:

* Any neurological condition that may place the subject at increased risk with exposure to botulinum toxin type A, including peripheral motor neuropathic diseases such as amyotrophic lateral sclerosis and motor neuropathy, and neuromuscular junctional disorders such as Lambert-Eaton syndrome and myasthenia gravis
* Active skin disease, infections or inflammation at the injection sites
* Plan to receive botulinum toxin type A anywhere in the face through the duration of the study
* History of allergy or sensitivity to any botulinum toxin preparations or to any component of the test article
* Current enrollment in an investigational drug or device trial or participation in such a trial within the last 30 days prior to screening through end of trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2016-12-08 (Actual); Primary Completion 2017-11-14 (Actual); Study Completion 2017-11-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Birmingham, Alabama
  - Beverly Hills, California
  - Newport Beach, California
  - San Francisco, California
  - Santa Monica, California
  - Greenwood, Colorado
  - Boca Raton, Florida
  - Coral Gables, Florida
  - Chestnut Hill, Massachusetts
  - Birmingham, Michigan
  - Montclair, New Jersey
  - New York, New York
  - Chapel Hill, North Carolina
  - Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bertucci V, Solish N, Kaufman-Janette J, Yoelin S, Shamban A, Schlessinger J, Snyder D, Gallagher C, Liu Y, Shears G, Rubio RG. DaxibotulinumtoxinA for Injection has a prolonged duration of response in the treatment of glabellar lines: Pooled data from two multicenter, randomized, double-blind, placebo-controlled, phase 3 studies (SAKURA 1 and SAKURA 2). J Am Acad Dermatol. 2020 Apr;82(4):838-845. doi: 10.1016/j.jaad.2019.06.1313. Epub 2019 Nov 29. PMID 31791824
- [Derived] Carruthers JD, Fagien S, Joseph JH, Humphrey SD, Biesman BS, Gallagher CJ, Liu Y, Rubio RG; SAKURA 1 and SAKURA 2 Investigator Group; SAKURA 1 and SAKURA 2 Investigator Group includes the following. DaxibotulinumtoxinA for Injection for the Treatment of Glabellar Lines: Results from Each of Two Multicenter, Randomized, Double-Blind, Placebo-Controlled, Phase 3 Studies (SAKURA 1 and SAKURA 2). Plast Reconstr Surg. 2020 Jan;145(1):45-58. doi: 10.1097/PRS.0000000000006327. PMID 31609882

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Outpatient, male or non-pregnant, non-nursing females, 18-75 years of age, and in good general health with moderate (2) or severe (3) glabellar lines during maximum frown based on the IGA-FWS and PFWS.
Groups:
- Placebo: Biological/Vaccine: Placebo Intramuscular injection
  Placebo: Intramuscular injection
Period: Overall Study
Arm/Group | DaxibotulinumtoxinA 40 Units | Placebo
Started | 201 | 102
Completed | 182 | 93
Not Completed | 19 | 9

BASELINE CHARACTERISTICS:
Population: Intent to treat population
Groups:
- Total: Total of all reporting groups
Arm/Group | DaxibotulinumtoxinA 40 Units | Placebo | Total
Number analyzed (Participants) | 201 | 102 | 303
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 180 | 95 | 275
  >=65 years | 21 | 7 | 28
Age, Continuous [Mean (Full Range); unit: years] | 50.9 [23 to 74] | 49.0 [22 to 74] | 50.3 [22 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 174 | 88 | 262
  Male | 27 | 14 | 41
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 7 | 2 | 9
  Race: American Indian or Alaska Native American | 0 | 1 | 1
  Race: Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Race: Black of African American | 10 | 8 | 18
  Race: More than one race | 1 | 2 | 3
  Race: Unknown or Not Reported | 10 | 7 | 17
  Race: White | 173 | 81 | 254
Region of Enrollment [Number; unit: participants]
  United States | 201 | 102 | 303

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects Who Achieved ≥ 2 Point Improvement Independently and Concurrently on Investigator and Patient Rating Scales
Description: Percentage of subjects who achieve at least a 2-point improvement from baseline and a score of 0 or 1 (i.e., none or mild wrinkles in severity) on both Investigator and Subject Frown Wrinkle Severity (FWS) assessments
Time Frame: Week 4
Population: Intent to treat population
Measure: Number; unit: percentage of subjects
Groups:
- DaxibotulinumtoxinA: Biological/Vaccine: Botulinum Toxins, Type A Intramuscular injection
  Botulinum Toxins, Type A: Intramuscular injection
- Placebo: Biological/Vaccine: Placebo Intramuscular injection
  Placebos: Intramuscular injection
Arm/Group | DaxibotulinumtoxinA | Placebo
Number analyzed (Participants) | 201 | 102
percentage of subjects | 73.6 | 0

2. Secondary Outcome: The Time to Return to Moderate to Severe on Both IGA-FWS and PFWS Scales for DaxibotulinumtoxinA for Injection Group
Description: The duration of response will be evaluated by analyzing the number of days to return to moderate or severe on both IGA-FWS and PFWS scales for DaxibotulinumtoxinA for Injection group.
Time Frame: 0-36 weeks
Population: ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | DaxibotulinumtoxinA 40 Units
Number analyzed (Participants) | 201
days | 168 [164 to 169]

3. Secondary Outcome: The Time to Return to, or Worse Than, Baseline on Both IGA-FWS and PFWS Scales for DaxibotulinumtoxinA for Injection Group
Description: The duration of response will be evaluated by analyzing the number of days to return to, or worse than, baseline on both IGA-FWS and PFWS scales for DaxibotulinumtoxinA for Injection group.
Time Frame: 0-36 weeks
Population: ITT population
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | DaxibotulinumtoxinA 40 Units
Number analyzed (Participants) | 201
days | 194 [173 to 196]

ADVERSE EVENTS:
Time Frame: The adverse events were collected throughout the entire study, up to 36 weeks
Description: The Safety Population includes all subjects who received at least 1 study treatment injection and was used to assess AEs and SAEs.
Arm/Group | DaxibotulinumtoxinA 40 Units | Placebo
All-Cause Mortality (participants affected / at risk) | 0/201 | 0/102
Serious Adverse Events (participants affected / at risk) | 2/201 | 1/102
Other Adverse Events (participants affected / at risk) | 29/201 | 7/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DaxibotulinumtoxinA 40 Units (N=201) | Placebo (N=102)
Bone marrow failure (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DaxibotulinumtoxinA 40 Units (N=201) | Placebo (N=102)
Injection Site Pain (General disorders) | 10 (10) | 4 (4)
Headache (Nervous system disorders) | 19 (19) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
With respect to any proposed publication or disclosure of the results of the Study, the Study Center and Investigator shall submit to Revance a copy of the proposed publication or disclosure at least sixty (60) days prior to the submission thereof for publication or disclosure to a third party: (i) to provide Revance with the opportunity to review and comment on the contents thereof, and (ii) to identify any Confidential Information to be deleted from the proposed publication or disclosure.

DOCUMENTS (2):
  • Study Protocol (2016-11-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT03014622/Prot_000.pdf
  • Statistical Analysis Plan (2017-11-21): https://cdn.clinicaltrials.gov/large-docs/22/NCT03014622/SAP_001.pdf